CLINICAL TRIAL: NCT05457881
Title: Short-Term Endogenous Hydrogen Sulfide Upregulation For Vein Graft Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funds to start study
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, C. Keith Ozaki, M.D., F.A.C.S., John A. Mannick Professor of Surgery, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021P002206
Record Dates: First submitted 2022-02-07; First posted 2022-07-14 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Vascular Diseases; Surgery
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Intervention Model Description: 3:2 randomization to short-term protein calorie restriction diet versus regular meals prior to elective major vascular surgery
Who Masked: Investigator, Outcomes Assessor
Masking Description: Subjects will be discretely randomized by the clinical research assistants upon final clearance for their procedure by the anesthesiology service, and their assigned group will be concealed to all subsequent team members (clinicians, research scientists, statistician) until data lock
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein-calorie restriction (Experimental): Four day dietary intervention immediately before surgery of Scandi-Shake [any of 4 flavors - vanilla, strawberry, banana cream, and caramel] mixed with almond milk (85 grams Scandi-Shake mix to 240 cc almond milk) calculated individually for a total daily volume to achieve 30% caloric restriction and 70% protein restriction, based on gender, age, height, weight, and activity level.
  Interventions: Dietary Supplement: Scandi-Shake
- Control (No Intervention): Ad libitum diet for four days immediately before surgery

INTERVENTIONS:
Dietary Supplement: Scandi-Shake — Scandi-Shake [any of 4 flavors - vanilla, strawberry, banana cream, and caramel] mixed with almond milk (85 grams Scandi-Shake mix to 240 cc almond milk), calculated individually for a total daily volume to achieve 30% caloric restriction and 70% protein restriction, based on ideal body weight. The Mifflin St. Jeor equation will be used to calculate the total 24-hour energy needs based on gender, age, height, weight, and activity factor for the PCR diet. Daily physical activity will be assessed by questionnaire to determine the activity factor for accurate calorie restriction calculations. Nutritionists will use this equation to create a unique shake for each individual patient. The shakes will be separated into 4 equal portions per day, for a total of 16 portions across the 4 pre-operative days. Patients can consume the 4 daily portions at whichever time of day they choose. The shakes are frozen 24 hours before distribution.
  Arms: Protein-calorie restriction

SUMMARY:
A randomized, controlled trial to evaluate patient compliance and biologic mechanisms of a short-term pre-operative Protein-Calorie Restriction (PCR) diet in comparison to a normal ad libitum diet for 4 days before elective vascular surgery involving a major operation. After a pilot study exploring the safety and feasibility of the PCR diet conducted inpatient before carotid endarterectomy titled Short-Term Endogenous Hydrogen Sulfide Upregulation, and a follow-up study titled Dietary Restriction in Vascular Surgery, the investigators now aim to expand the study to at home diet among a variety of vascular surgery procedures. This study will further elucidate not only the practicality of pre-operative short term dietary restriction, but also provide early data to inform biologic mechanisms and to inform future efficacy trails.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) remains a major health issue in the United States, especially with the metabolic syndrome and aging population. Surgical bypass using autogenous vein remains the most effective and durable choice for patients with advanced PAD. However, these vascular interventions suffer from high failure rates due to the development of significant occlusive lesions (intimal hyperplasia [IH]). Similar failure mechanisms plague coronary artery bypass grafts and endovascular interventions. Despite decades of vein graft research, our understanding of the biologic mechanisms of vein graft failure remains obscure.

Hydrogen sulfide (H2S) has emerged as a critical gaseous signaling molecule in multiple processes including ischemia/reperfusion (IR) injury, angiogenesis, intimal hyperplasia, and anti-inflammatory mechanisms. It even appears to hold anti-atherosclerotic properties. However, the gas is toxic with a half-life of minutes, and it can be rapidly oxidized. Furthermore, clinically useful pharmacologic H2S donors have not been developed to date. In our 2015 Cell paper the investigators link substantial upregulation of endogenous H2S via short-term manipulation of mammalian dietary intake: simple dietary restriction. Our first pilot study had aims to determine the feasibility and safety of a PCR diet in vascular patients, concluding with no significant serious adverse events in any of the patients receiving the diet. The investigators learned that patients do not like having to stay in the hospital research unit pre-operatively. Long term the investigators aim to substantively impact the vascular patient at several levels: protection from IR, intimal hyperplasia, peri-procedural events such as stroke, cardiac dysfunction and myocardial infarction, and promotion of angiogenesis. For the current effort, the investigators will focus on potential biologic mechanisms of PCR and feasibility of eventual larger initiatives to accomplish this long-term aim.

A powerful method to upregulate H2S is PCR. Defined as reduced food intake without malnutrition, PCR is best known for extending lifespan in model organisms from yeast to non-human primates. The efficacy of PCR against acute stress, including surgical stress, in preclinical models is also well established. Pilot studies suggest that humans respond to PCR in beneficial ways with respect to metabolic fitness (including improved glucose homeostasis, lipid profiles, and cardiovascular performance). But humans also have great difficulty complying with long-term voluntary food restriction, which is a prime reason that PCR has not been previously exploited in the clinical setting despite promising efficacy. However, recent data in model organisms point to a rapid onset of PCR benefits and challenges the notion that long-term PCR is required for benefits to accrue. In fruit flies, the maximal benefit of PCR on mortality risk occurs within 2-3 days. In rodents, the investigators have shown that surgical stress resistance also occurs within days, and the benefits center on upregulation of endogenous H2S. Nonetheless, except for pre-operative overnight fasting (which serves a different purpose) dietary recommendations are largely absent from peri-op management.

Pilot data suggest that adverse post-operative outcomes linked to oxidative stress, inflammation and stress hormones may be modified by brief PCR in humans as well. In subjects who undertook food restriction for 12 hours per day for a month, markers of inflammation decreased significantly. PCR has been shown to reduce oxidative stress in both chronic and acute settings. Similarly, PCR may decrease stress hormone release. PCR also appears to work rapidly even in obese individuals or ill individuals. In gastric bypass surgery, two weeks of PCR reduced the risk of complications and procedure difficulty. With respect to patient compliance, brief (4 days to 2 weeks) pre-operative dietary interventions have been shown to be feasible and safe in selected patients, ranging from obese candidates for laparoscopic surgery to living organ donors. In our own human pilot research, vascular surgery patients have safely completed 3 days of pre-operative PCR diet without serious adverse events or reactions.

For the current project the investigators propose a randomized, controlled trial to evaluate patient compliance and biologic effects of a short-term pre-operative PCR diet in comparison to a normal ad libitum diet for 4 days before elective vascular surgery involving an open major operation. This mechanistic clinical study is structured as a prospective, multi-year study of 226 vascular surgery patients undergoing non-emergency lower-extremity arterial vein bypass surgery randomized into two pre-operative dietary groups: observational group (n=90) and PCR (commercially available ScandiShake x 4 days, n=136). This specific dietary intervention to upregulate endogenous H2S is based on our preliminary data balanced with economic and clinical feasibility considerations. The event rate for the control group is assumed to be 33% based on the literature and data largely from our institutions. Our goal is to find a suitable (total) sample size for power 1 - β=0.8 at 5% level of significance. It has been assumed that Relative Risk Reduction (RRR) is 50% or Absolute Risk Reduction (ARR) is 16.5%. Projected total sample size, for treatment group to control group ratio of 1.5 (60% to 40%), is 225.55 which approximate to 226. For the structure of our dietary intervention this means 90 for the control group and 136 for the treatment group. However, it must be emphasized that the primary goal of this project is to decipher mechanisms in humans rather than evaluate clinical efficacy.

Employing this randomized (3:2), parallel design, subjects will be assigned to either the supervised PCR diet (Scandi-Shake [any of 4 flavors - vanilla, strawberry, banana cream, and caramel] mixed with almond milk (85 grams Scandi-Shake mix to 240 cc almond milk), calculated individually for a total daily volume to achieve 30% caloric restriction and 70% protein restriction, based on ideal body weight), or continued routine ad libitum diet. The Mifflin St.Jeor equation will be used to calculate the total 24-hour energy needs based on gender, age, height, weight, and activity factor for the PCR diet. Daily physical activity will be assessed by questionnaire to determine the activity factor for accurate calorie restriction calculations. Nutritionists will use this equation to create a unique shake for each individual patient. The entire course of the dietary intervention will occur only during the 4 days prior to surgery. The shakes will be separated into 4 equal portions per day, for a total of 16 portions across the 4 pre-operative days. Patients can consume the 4 daily portions at whichever time of day they choose. The shakes are frozen 24 hours before distribution. Water intake is ad libitum for both cohorts.

Subjects will be discretely randomized by the clinical research assistants upon final clearance for their procedure by the anesthesiology service, and their assigned group will be concealed to all subsequent team members (clinicians, research scientists, statistician) until data lock. Subjects in both cohorts will log their diet in the mobile application MealLogger. This app allows the subject to post a photo and short description of their food from a mobile device and directly share the information with the study coordinator. Staff can communicate through the app with subjects to clarify what exactly was eaten.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients planned for non-emergency lower extremity vein bypass surgery
* Projected survival of at least one year
* Ability to provide informed consent
* Albumin ≥3.0 and negative pregnancy test (if relevant)
* No known allergy to Scandi-Shake ingredients

Exclusion Criteria:

* <18 years of age
* Emergency lower extremity vascular surgery
* Projected survival of < one year
* Albumin <3.0
* Pregnancy, intention to become pregnant, or lack of standard contraception method
* Allergy to Scandi-Shake ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Compliance with outpatient Protein-Calorie Restriction measured via food diary | 1 Month
  Subject compliance with PCR will be measured through direct dietary intake data via food diary in comparison to the ad libitum diet. But one of the indirect goals of the initiative is to better understand how compliance can be assessed in this population.
Compliance with outpatient Protein-Calorie Restriction measured via biologic assays for plasma free amino acids | 1 Month
  Subject compliance with PCR will be measured through biologic assays (e.g., plasma free amino acids) in comparison to the ad libitum diet. But one of the indirect goals of the initiative is to better understand how compliance can be assessed in this population.
Compliance with outpatient Protein-Calorie Restriction measured via biologic assays for pre-albumin | 1 Month
  Subject compliance with PCR will be measured through biologic assays (e.g., insulin-like growth factor) in comparison to the ad libitum diet. But one of the indirect goals of the initiative is to better understand how compliance can be assessed in this population.
Compliance with outpatient Protein-Calorie Restriction measured via biologic assays insulin-like growth factor | 1 Month
  Subject compliance with PCR will be measured through direct dietary intake data via food diary, and we will also have biologic assays for serum markers including plasma free amino acids, pre-albumin, and insulin-like growth factor in comparison to the ad libitum diet. But, one of the indirect goals of the initiative is to better understand how compliance can be assessed in this population.
Change over time from baseline values to values before surgery and day 1 after surgery in the comparison of H2S and standard biological markers of stress in blood | Baseline, Day 0, Day 1
  H2S and standard biological markers of stress are collected at baseline, immediately before surgery, and day 1 after surgery. Biological markers include: adipose phenotyping (quantification of adipokines, adipose derived hormones), leukocyte phenotyping and quantification via flow cytometry, and serum assays of IL-1beta, IL-6, IL-8, HGF, leptin, MCP-1, PAI-1, resistin, NGF, TNF, adiponectin, hydrogen sulfide (including production capacity) assays, insulin, lipid panels, FGF 21, pre-albumin, epinephrine, norepinephrine, dopamine, CBC with differential, basic metabolic panel including calcium. These biomarkers will be quantified in the various tissues for individual participants and be mathematically aggregated for groups (i.e., an aggregate unit of measurement will be used)"
Major Adverse Limb Event | 2 years
  Untreated loss of conduit patency and/or severe limb ischemia leading to an intervention or major amputation. Includes acute limb ischemia (including the need for thrombectomy/ thrombolysis), major amputation (above the ankle), need for re-do surgical revascularization for the index limb.

SECONDARY OUTCOMES:
Comparison of surgical and medical complications | 1 Month
  These endpoints will include surgical and medical complications such as cardiac, neurologic, infectious, vascular, wound, and any other clinically significant events that occur within 30 days of surgery
One-year survival | 1 year
  Patient survival after one-year participating in the trial
Renal dysfunction, stroke, myocardial infarction, patency of the vein graft (primary, primary assisted, secondary), survival. | 1 Month, 1 year
  Medical record derived complications (using standardized NSQIP definitions and outcomes) +/- PCR. eGFR will be the primary measure of renal function.
  These data will be integrated mathematically to combine all the features in an additive model to develop the final integrative model.
Wound Complication | 1 Month
  Superficial Surgical Site Infection (SSI): Infection that involves only skin/ SQ tissue of the incision and at least one of the following: Purulent drainage, Positive wound culture, At least one of the following signs/symptoms of infection: pain or tenderness, localized swelling, redness, or heat AND superficial incision is deliberately opened by the surgeon, unless incision is culture-negative, Diagnosis of superficial SSI by attending Deep SSI: Infection involves deep tissues (fascial/ muscle layers) of the incision and at least one of the following: Purulent drainage from the deep incision, A deep incision spontaneously dehisces or is deliberately opened by a surgeon when the patient has at least one of the following signs or symptoms: fever (> 38C), localized pain, or tenderness, unless site is culture-negative, An abscess or other evidence of infection involving the deep incision, Diagnosis of deep SSI by attending Dehiscence: Skin separation requiring local wound care.

OTHER OUTCOMES:
Gut microbiome Analysis | 0-34 days
  Through this analysis, we aim to:
  1. Delineate the vascular surgery patient gut microbiome baseline and in response to surgery +/- PCR and
  2. Define the impact of surgery (trauma, peri-procedural antibiotics, hospitalization, etc.) on the colonic microbiome, and the interplay of pre-operative PCR on these dynamics.
  For the gut microbiome analyses, stool samples will be collected and assayed via commercially available kits.
  Stool samples will be collected at baseline, day 1 of diet, day 2 of diet, day 3 of diet, day 4 of diet, the day of surgery, post-operative day 1, 14, and post-operative day 30
Microbiome-derived circulating metabolites | 0-34 days
  Specific Aim 2: Determine baseline active microbiome derived circulating metabolites in this cohort and measure the impact of PCR and surgery on these mediators.
  Specific Aim 2 Hypothesis: Short-term PCR in vascular surgery patients alters human gut origin circulating metabolites to a more favorable, metabolically protective phenotype
  Plasma will be sampled at baseline, the day of surgery, post-operative day 1, and post-operative day 30. Short chain fatty acids [SCFA] (acetate, butyrate, and propionate) will be quantified using liquid chromatography-tandem mass spectrometry. Indole- and phenyl-derived metabolites, including indole, serotonin, kynurenine, tryptophan, indole-3-propionic acid, indole-3-aldehyde, indoxyl sulfate, 3-hydroxyanthranilic acid, p-cresyl sulfate, and hippuric acid, will be additionally quantified using the previously described high-performance liquid chromatography and tandem mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Charles K Ozaki, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):e28-e292. doi: 10.1161/01.cir.0000441139.02102.80. Epub 2013 Dec 18. No abstract available. PMID 24352519
- [Background] Kraiss LW, Conte MS, Geary RL, Kibbe M, Ozaki CK. Setting high-impact clinical research priorities for the Society for Vascular Surgery. J Vasc Surg. 2013 Feb;57(2):493-500. doi: 10.1016/j.jvs.2012.09.069. PMID 23337859
- [Background] Adam DJ, Beard JD, Cleveland T, Bell J, Bradbury AW, Forbes JF, Fowkes FG, Gillepsie I, Ruckley CV, Raab G, Storkey H; BASIL trial participants. Bypass versus angioplasty in severe ischaemia of the leg (BASIL): multicentre, randomised controlled trial. Lancet. 2005 Dec 3;366(9501):1925-34. doi: 10.1016/S0140-6736(05)67704-5. PMID 16325694
- [Background] Bradbury AW. Bypass versus angioplasty in severe ischaemia of the leg (BASIL) trial: what are its implications? Semin Vasc Surg. 2009 Dec;22(4):267-74. doi: 10.1053/j.semvascsurg.2009.10.010. PMID 20006808
- [Background] Bradbury AW; BASIL trial Investigators and Participants. Bypass versus Angioplasty in Severe Ischaemia of the Leg (BASIL) trial in perspective. J Vasc Surg. 2010 May;51(5 Suppl):1S-4S. doi: 10.1016/j.jvs.2010.02.002. No abstract available. PMID 20435257
- [Background] Forbes JF, Adam DJ, Bell J, Fowkes FG, Gillespie I, Raab GM, Ruckley CV, Bradbury AW; BASIL trial Participants. Bypass versus Angioplasty in Severe Ischaemia of the Leg (BASIL) trial: Health-related quality of life outcomes, resource utilization, and cost-effectiveness analysis. J Vasc Surg. 2010 May;51(5 Suppl):43S-51S. doi: 10.1016/j.jvs.2010.01.076. PMID 20435261
- [Background] Bradbury AW, Adam DJ, Bell J, Forbes JF, Fowkes FG, Gillespie I, Raab G, Ruckley CV. Multicentre randomised controlled trial of the clinical and cost-effectiveness of a bypass-surgery-first versus a balloon-angioplasty-first revascularisation strategy for severe limb ischaemia due to infrainguinal disease. The Bypass versus Angioplasty in Severe Ischaemia of the Leg (BASIL) trial. Health Technol Assess. 2010 Mar;14(14):1-210, iii-iv. doi: 10.3310/hta14140. PMID 20307380
- [Background] Bradbury AW, Adam DJ, Bell J, Forbes JF, Fowkes FG, Gillespie I, Ruckley CV, Raab GM; BASIL trial Participants. Bypass versus Angioplasty in Severe Ischaemia of the Leg (BASIL) trial: An intention-to-treat analysis of amputation-free and overall survival in patients randomized to a bypass surgery-first or a balloon angioplasty-first revascularization strategy. J Vasc Surg. 2010 May;51(5 Suppl):5S-17S. doi: 10.1016/j.jvs.2010.01.073. PMID 20435258
- [Background] Conte MS, Bandyk DF, Clowes AW, Moneta GL, Seely L, Lorenz TJ, Namini H, Hamdan AD, Roddy SP, Belkin M, Berceli SA, DeMasi RJ, Samson RH, Berman SS; PREVENT III Investigators. Results of PREVENT III: a multicenter, randomized trial of edifoligide for the prevention of vein graft failure in lower extremity bypass surgery. J Vasc Surg. 2006 Apr;43(4):742-751; discussion 751. doi: 10.1016/j.jvs.2005.12.058. PMID 16616230
- [Background] Ozaki CK. Cytokines and the early vein graft: strategies to enhance durability. J Vasc Surg. 2007 Jun;45 Suppl A(Suppl A):A92-8. doi: 10.1016/j.jvs.2007.02.032. PMID 17544029
- [Background] Conte MS. Technical factors in lower-extremity vein bypass surgery: how can we improve outcomes? Semin Vasc Surg. 2009 Dec;22(4):227-33. doi: 10.1053/j.semvascsurg.2009.10.004. PMID 20006802
- [Background] Conte MS, Bandyk DF, Clowes AW, Moneta GL, Namini H, Seely L. Risk factors, medical therapies and perioperative events in limb salvage surgery: observations from the PREVENT III multicenter trial. J Vasc Surg. 2005 Sep;42(3):456-64; discussion 464-5. doi: 10.1016/j.jvs.2005.05.001. PMID 16171587
- [Background] Conte MS, Mann MJ, Simosa HF, Rhynhart KK, Mulligan RC. Genetic interventions for vein bypass graft disease: a review. J Vasc Surg. 2002 Nov;36(5):1040-52. doi: 10.1067/mva.2002.129112. PMID 12422116
- [Background] Schleifenbaum J, Kohn C, Voblova N, Dubrovska G, Zavarirskaya O, Gloe T, Crean CS, Luft FC, Huang Y, Schubert R, Gollasch M. Systemic peripheral artery relaxation by KCNQ channel openers and hydrogen sulfide. J Hypertens. 2010 Sep;28(9):1875-82. doi: 10.1097/HJH.0b013e32833c20d5. PMID 20577128
- [Background] Polhemus D, Kondo K, Bhushan S, Bir SC, Kevil CG, Murohara T, Lefer DJ, Calvert JW. Hydrogen sulfide attenuates cardiac dysfunction after heart failure via induction of angiogenesis. Circ Heart Fail. 2013 Sep 1;6(5):1077-86. doi: 10.1161/CIRCHEARTFAILURE.113.000299. Epub 2013 Jun 28. PMID 23811964
- [Background] Kondo K, Bhushan S, King AL, Prabhu SD, Hamid T, Koenig S, Murohara T, Predmore BL, Gojon G Sr, Gojon G Jr, Wang R, Karusula N, Nicholson CK, Calvert JW, Lefer DJ. H(2)S protects against pressure overload-induced heart failure via upregulation of endothelial nitric oxide synthase. Circulation. 2013 Mar 12;127(10):1116-27. doi: 10.1161/CIRCULATIONAHA.112.000855. Epub 2013 Feb 7. PMID 23393010
- [Background] Hine C, Mitchell JR. Calorie restriction and methionine restriction in control of endogenous hydrogen sulfide production by the transsulfuration pathway. Exp Gerontol. 2015 Aug;68:26-32. doi: 10.1016/j.exger.2014.12.010. Epub 2014 Dec 16. PMID 25523462
- [Background] King AL, Polhemus DJ, Bhushan S, Otsuka H, Kondo K, Nicholson CK, Bradley JM, Islam KN, Calvert JW, Tao YX, Dugas TR, Kelley EE, Elrod JW, Huang PL, Wang R, Lefer DJ. Hydrogen sulfide cytoprotective signaling is endothelial nitric oxide synthase-nitric oxide dependent. Proc Natl Acad Sci U S A. 2014 Feb 25;111(8):3182-7. doi: 10.1073/pnas.1321871111. Epub 2014 Feb 10. PMID 24516168
- [Background] Hine C, Harputlugil E, Zhang Y, Ruckenstuhl C, Lee BC, Brace L, Longchamp A, Trevino-Villarreal JH, Mejia P, Ozaki CK, Wang R, Gladyshev VN, Madeo F, Mair WB, Mitchell JR. Endogenous hydrogen sulfide production is essential for dietary restriction benefits. Cell. 2015 Jan 15;160(1-2):132-44. doi: 10.1016/j.cell.2014.11.048. Epub 2014 Dec 23. PMID 25542313
- [Background] Xie L, Gu Y, Wen M, Zhao S, Wang W, Ma Y, Meng G, Han Y, Wang Y, Liu G, Moore PK, Wang X, Wang H, Zhang Z, Yu Y, Ferro A, Huang Z, Ji Y. Hydrogen Sulfide Induces Keap1 S-sulfhydration and Suppresses Diabetes-Accelerated Atherosclerosis via Nrf2 Activation. Diabetes. 2016 Oct;65(10):3171-84. doi: 10.2337/db16-0020. Epub 2016 Jun 22. PMID 27335232
- [Background] Longchamp A, Mirabella T, Arduini A, MacArthur MR, Das A, Trevino-Villarreal JH, Hine C, Ben-Sahra I, Knudsen NH, Brace LE, Reynolds J, Mejia P, Tao M, Sharma G, Wang R, Corpataux JM, Haefliger JA, Ahn KH, Lee CH, Manning BD, Sinclair DA, Chen CS, Ozaki CK, Mitchell JR. Amino Acid Restriction Triggers Angiogenesis via GCN2/ATF4 Regulation of VEGF and H2S Production. Cell. 2018 Mar 22;173(1):117-129.e14. doi: 10.1016/j.cell.2018.03.001. PMID 29570992
- [Background] Harputlugil E, Hine C, Vargas D, Robertson L, Manning BD, Mitchell JR. The TSC complex is required for the benefits of dietary protein restriction on stress resistance in vivo. Cell Rep. 2014 Aug 21;8(4):1160-70. doi: 10.1016/j.celrep.2014.07.018. Epub 2014 Aug 14. PMID 25131199
- [Background] Robertson LT, Trevino-Villarreal JH, Mejia P, Grondin Y, Harputlugil E, Hine C, Vargas D, Zheng H, Ozaki CK, Kristal BS, Simpson SJ, Mitchell JR. Protein and Calorie Restriction Contribute Additively to Protection from Renal Ischemia Reperfusion Injury Partly via Leptin Reduction in Male Mice. J Nutr. 2015 Aug;145(8):1717-27. doi: 10.3945/jn.114.199380. Epub 2015 Jun 3. PMID 26041674
- [Background] Mitchell JR, Beckman JA, Nguyen LL, Ozaki CK. Reducing elective vascular surgery perioperative risk with brief preoperative dietary restriction. Surgery. 2013 Apr;153(4):594-8. doi: 10.1016/j.surg.2012.09.007. Epub 2012 Dec 4. PMID 23218877
- [Background] Nguyen B, Tao M, Yu P, Mauro C, Seidman MA, Wang YE, Mitchell J, Ozaki CK. Preoperative diet impacts the adipose tissue response to surgical trauma. Surgery. 2013 Apr;153(4):584-93. doi: 10.1016/j.surg.2012.11.001. Epub 2012 Dec 27. PMID 23274098
- [Background] Mauro CR, Tao M, Yu P, Trevino-Villerreal JH, Longchamp A, Kristal BS, Ozaki CK, Mitchell JR. Preoperative dietary restriction reduces intimal hyperplasia and protects from ischemia-reperfusion injury. J Vasc Surg. 2016 Feb;63(2):500-9.e1. doi: 10.1016/j.jvs.2014.07.004. Epub 2014 Aug 8. PMID 25124359
- [Background] Kip P, Tao M, Trocha KM, MacArthur MR, Peters HAB, Mitchell SJ, Mann CG, Sluiter TJ, Jung J, Patterson S, Quax PHA, de Vries MR, Mitchell JR, Keith Ozaki C. Periprocedural Hydrogen Sulfide Therapy Improves Vascular Remodeling and Attenuates Vein Graft Disease. J Am Heart Assoc. 2020 Nov 17;9(22):e016391. doi: 10.1161/JAHA.120.016391. Epub 2020 Nov 4. PMID 33146045
- [Background] Maeda H, Gleiser CA, Masoro EJ, Murata I, McMahan CA, Yu BP. Nutritional influences on aging of Fischer 344 rats: II. Pathology. J Gerontol. 1985 Nov;40(6):671-88. doi: 10.1093/geronj/40.6.671. PMID 4056322
- [Background] Fontana L, Partridge L, Longo VD. Extending healthy life span--from yeast to humans. Science. 2010 Apr 16;328(5976):321-6. doi: 10.1126/science.1172539. PMID 20395504
- [Background] Mitchell JR, Verweij M, Brand K, van de Ven M, Goemaere N, van den Engel S, Chu T, Forrer F, Muller C, de Jong M, van IJcken W, IJzermans JN, Hoeijmakers JH, de Bruin RW. Short-term dietary restriction and fasting precondition against ischemia reperfusion injury in mice. Aging Cell. 2010 Feb;9(1):40-53. doi: 10.1111/j.1474-9726.2009.00532.x. Epub 2009 Oct 30. PMID 19878145
- [Background] van Ginhoven TM, Dik WA, Mitchell JR, Smits-te Nijenhuis MA, van Holten-Neelen C, Hooijkaas H, Hoeijmakers JH, de Bruin RW, IJzermans JN. Dietary restriction modifies certain aspects of the postoperative acute phase response. J Surg Res. 2011 Dec;171(2):582-9. doi: 10.1016/j.jss.2010.03.038. Epub 2010 Apr 13. PMID 20538300
- [Background] Speakman JR, Mitchell SE. Caloric restriction. Mol Aspects Med. 2011 Jun;32(3):159-221. doi: 10.1016/j.mam.2011.07.001. Epub 2011 Aug 10. PMID 21840335
- [Background] Longo VD, Mattson MP. Fasting: molecular mechanisms and clinical applications. Cell Metab. 2014 Feb 4;19(2):181-92. doi: 10.1016/j.cmet.2013.12.008. Epub 2014 Jan 16. PMID 24440038
- [Background] Varendi K, Airavaara M, Anttila J, Vose S, Planken A, Saarma M, Mitchell JR, Andressoo JO. Short-term preoperative dietary restriction is neuroprotective in a rat focal stroke model. PLoS One. 2014 Apr 4;9(4):e93911. doi: 10.1371/journal.pone.0093911. eCollection 2014. PMID 24705386
- [Background] Mejia P, Trevino-Villarreal JH, Hine C, Harputlugil E, Lang S, Calay E, Rogers R, Wirth D, Duraisingh MT, Mitchell JR. Dietary restriction protects against experimental cerebral malaria via leptin modulation and T-cell mTORC1 suppression. Nat Commun. 2015 Jan 30;6:6050. doi: 10.1038/ncomms7050. PMID 25636003
- [Background] Kip P, Trocha KM, Tao M, O'leary JJ, Ruske J, Giulietti JM, Trevino-Villareal JH, MacArthur MR, Bolze A, Burak MF, Patterson S, Ho KJ, Carmody RN, Guzman RJ, Mitchell JR, Ozaki CK. Insights From a Short-Term Protein-Calorie Restriction Exploratory Trial in Elective Carotid Endarterectomy Patients. Vasc Endovascular Surg. 2019 Aug;53(6):470-476. doi: 10.1177/1538574419856453. Epub 2019 Jun 19. PMID 31216949
- [Background] Glagov S. Intimal hyperplasia, vascular modeling, and the restenosis problem. Circulation. 1994 Jun;89(6):2888-91. doi: 10.1161/01.cir.89.6.2888. No abstract available. PMID 8205705
- [Background] Newby AC, Zaltsman AB. Molecular mechanisms in intimal hyperplasia. J Pathol. 2000 Feb;190(3):300-9. doi: 10.1002/(SICI)1096-9896(200002)190:33.0.CO;2-I. PMID 10685064
- [Background] Wu J, Zhang C. Neointimal hyperplasia, vein graft remodeling, and long-term patency. Am J Physiol Heart Circ Physiol. 2009 Oct;297(4):H1194-5. doi: 10.1152/ajpheart.00703.2009. Epub 2009 Aug 7. No abstract available. PMID 19666837
- [Background] Chiu JJ, Chien S. Effects of disturbed flow on vascular endothelium: pathophysiological basis and clinical perspectives. Physiol Rev. 2011 Jan;91(1):327-87. doi: 10.1152/physrev.00047.2009. PMID 21248169
- [Background] Berceli SA, Davies MG, Kenagy RD, Clowes AW. Flow-induced neointimal regression in baboon polytetrafluoroethylene grafts is associated with decreased cell proliferation and increased apoptosis. J Vasc Surg. 2002 Dec;36(6):1248-55. doi: 10.1067/mva.2002.128295. PMID 12469058
- [Background] Jiang Z, Wu L, Miller BL, Goldman DR, Fernandez CM, Abouhamze ZS, Ozaki CK, Berceli SA. A novel vein graft model: adaptation to differential flow environments. Am J Physiol Heart Circ Physiol. 2004 Jan;286(1):H240-5. doi: 10.1152/ajpheart.00760.2003. Epub 2003 Sep 18. PMID 14500133
- [Background] Lal BK, Beach KW, Roubin GS, Lutsep HL, Moore WS, Malas MB, Chiu D, Gonzales NR, Burke JL, Rinaldi M, Elmore JR, Weaver FA, Narins CR, Foster M, Hodgson KJ, Shepard AD, Meschia JF, Bergelin RO, Voeks JH, Howard G, Brott TG; CREST Investigators. Restenosis after carotid artery stenting and endarterectomy: a secondary analysis of CREST, a randomised controlled trial. Lancet Neurol. 2012 Sep;11(9):755-63. doi: 10.1016/S1474-4422(12)70159-X. Epub 2012 Aug 2. PMID 22857850
- [Background] Alexander JH, Hafley G, Harrington RA, Peterson ED, Ferguson TB Jr, Lorenz TJ, Goyal A, Gibson M, Mack MJ, Gennevois D, Califf RM, Kouchoukos NT; PREVENT IV Investigators. Efficacy and safety of edifoligide, an E2F transcription factor decoy, for prevention of vein graft failure following coronary artery bypass graft surgery: PREVENT IV: a randomized controlled trial. JAMA. 2005 Nov 16;294(19):2446-54. doi: 10.1001/jama.294.19.2446. PMID 16287955
- [Background] Dember LM, Beck GJ, Allon M, Delmez JA, Dixon BS, Greenberg A, Himmelfarb J, Vazquez MA, Gassman JJ, Greene T, Radeva MK, Braden GL, Ikizler TA, Rocco MV, Davidson IJ, Kaufman JS, Meyers CM, Kusek JW, Feldman HI; Dialysis Access Consortium Study Group. Effect of clopidogrel on early failure of arteriovenous fistulas for hemodialysis: a randomized controlled trial. JAMA. 2008 May 14;299(18):2164-71. doi: 10.1001/jama.299.18.2164. PMID 18477783
- [Background] Beathard GA, Arnold P, Jackson J, Litchfield T; Physician Operators Forum of RMS Lifeline. Aggressive treatment of early fistula failure. Kidney Int. 2003 Oct;64(4):1487-94. doi: 10.1046/j.1523-1755.2003.00210.x. PMID 12969170
- [Background] Lee T, Roy-Chaudhury P. Advances and new frontiers in the pathophysiology of venous neointimal hyperplasia and dialysis access stenosis. Adv Chronic Kidney Dis. 2009 Sep;16(5):329-38. doi: 10.1053/j.ackd.2009.06.009. PMID 19695501
- [Background] Grondin CM, Meere C, Castonguay Y, Lepage G, Grondin P. Progressive and late obstruction of an aorto-coronary venous bypass graft. Circulation. 1971 May;43(5):698-702. doi: 10.1161/01.cir.43.5.698. No abstract available. PMID 5578845
- [Background] Davies MG, Hagen PO. Pathophysiology of vein graft failure: a review. Eur J Vasc Endovasc Surg. 1995 Jan;9(1):7-18. doi: 10.1016/s1078-5884(05)80218-7. PMID 7664016
- [Background] Lemson MS, Tordoir JH, Daemen MJ, Kitslaar PJ. Intimal hyperplasia in vascular grafts. Eur J Vasc Endovasc Surg. 2000 Apr;19(4):336-50. doi: 10.1053/ejvs.1999.1040. No abstract available. PMID 10801366
- [Background] Subbotin VM. Analysis of arterial intimal hyperplasia: review and hypothesis. Theor Biol Med Model. 2007 Oct 31;4:41. doi: 10.1186/1742-4682-4-41. PMID 17974015
- [Background] Berceli SA, Jiang Z, Klingman NV, Pfahnl CL, Abouhamze ZS, Frase CD, Schultz GS, Ozaki CK. Differential expression and activity of matrix metalloproteinases during flow-modulated vein graft remodeling. J Vasc Surg. 2004 May;39(5):1084-90. doi: 10.1016/j.jvs.2003.12.031. PMID 15111865
- [Background] Berceli SA, Jiang Z, Klingman NV, Schultz GS, Ozaki CK. Early differential MMP-2 and -9 dynamics during flow-induced arterial and vein graft adaptations. J Surg Res. 2006 Aug;134(2):327-34. doi: 10.1016/j.jss.2005.12.030. Epub 2006 Feb 20. PMID 16488440
- [Background] Rectenwald JE, Moldawer LL, Huber TS, Seeger JM, Ozaki CK. Direct evidence for cytokine involvement in neointimal hyperplasia. Circulation. 2000 Oct 3;102(14):1697-702. doi: 10.1161/01.cir.102.14.1697. PMID 11015350
- [Background] Jiang Z, Berceli SA, Pfahnl CL, Wu L, Goldman D, Tao M, Kagayama M, Matsukawa A, Ozaki CK. Wall shear modulation of cytokines in early vein grafts. J Vasc Surg. 2004 Aug;40(2):345-50. doi: 10.1016/j.jvs.2004.03.048. PMID 15297832
- [Background] Jiang Z, Shukla A, Miller BL, Espino DR, Tao M, Berceli SA, Ozaki CK. Tumor necrosis factor-alpha and the early vein graft. J Vasc Surg. 2007 Jan;45(1):169-76. doi: 10.1016/j.jvs.2006.08.049. PMID 17210403
- [Background] Colman RJ, Anderson RM, Johnson SC, Kastman EK, Kosmatka KJ, Beasley TM, Allison DB, Cruzen C, Simmons HA, Kemnitz JW, Weindruch R. Caloric restriction delays disease onset and mortality in rhesus monkeys. Science. 2009 Jul 10;325(5937):201-4. doi: 10.1126/science.1173635. PMID 19590001
- [Background] Richardson A, Liu F, Adamo ML, Van Remmen H, Nelson JF. The role of insulin and insulin-like growth factor-I in mammalian ageing. Best Pract Res Clin Endocrinol Metab. 2004 Sep;18(3):393-406. doi: 10.1016/j.beem.2004.02.002. PMID 15261845
- [Background] Shinmura K, Tamaki K, Bolli R. Impact of 6-mo caloric restriction on myocardial ischemic tolerance: possible involvement of nitric oxide-dependent increase in nuclear Sirt1. Am J Physiol Heart Circ Physiol. 2008 Dec;295(6):H2348-55. doi: 10.1152/ajpheart.00602.2008. Epub 2008 Oct 17. PMID 18931029
- [Background] Shinmura K, Tamaki K, Saito K, Nakano Y, Tobe T, Bolli R. Cardioprotective effects of short-term caloric restriction are mediated by adiponectin via activation of AMP-activated protein kinase. Circulation. 2007 Dec 11;116(24):2809-17. doi: 10.1161/CIRCULATIONAHA.107.725697. Epub 2007 Nov 26. PMID 18040027
- [Background] Chandrasekar B, Nelson JF, Colston JT, Freeman GL. Calorie restriction attenuates inflammatory responses to myocardial ischemia-reperfusion injury. Am J Physiol Heart Circ Physiol. 2001 May;280(5):H2094-102. doi: 10.1152/ajpheart.2001.280.5.H2094. PMID 11299211
- [Background] Yu ZF, Mattson MP. Dietary restriction and 2-deoxyglucose administration reduce focal ischemic brain damage and improve behavioral outcome: evidence for a preconditioning mechanism. J Neurosci Res. 1999 Sep 15;57(6):830-9. PMID 10467254
- [Background] Ahmet I, Wan R, Mattson MP, Lakatta EG, Talan M. Cardioprotection by intermittent fasting in rats. Circulation. 2005 Nov 15;112(20):3115-21. doi: 10.1161/CIRCULATIONAHA.105.563817. Epub 2005 Nov 7. PMID 16275865
- [Background] Heilbronn LK, Smith SR, Martin CK, Anton SD, Ravussin E. Alternate-day fasting in nonobese subjects: effects on body weight, body composition, and energy metabolism. Am J Clin Nutr. 2005 Jan;81(1):69-73. doi: 10.1093/ajcn/81.1.69. PMID 15640462
- [Background] Trepanowski JF, Canale RE, Marshall KE, Kabir MM, Bloomer RJ. Impact of caloric and dietary restriction regimens on markers of health and longevity in humans and animals: a summary of available findings. Nutr J. 2011 Oct 7;10:107. doi: 10.1186/1475-2891-10-107. PMID 21981968
- [Background] Cheng CW, Villani V, Buono R, Wei M, Kumar S, Yilmaz OH, Cohen P, Sneddon JB, Perin L, Longo VD. Fasting-Mimicking Diet Promotes Ngn3-Driven beta-Cell Regeneration to Reverse Diabetes. Cell. 2017 Feb 23;168(5):775-788.e12. doi: 10.1016/j.cell.2017.01.040. PMID 28235195
- [Background] Mair W, Goymer P, Pletcher SD, Partridge L. Demography of dietary restriction and death in Drosophila. Science. 2003 Sep 19;301(5640):1731-3. doi: 10.1126/science.1086016. PMID 14500985
- [Background] Peng W, Robertson L, Gallinetti J, Mejia P, Vose S, Charlip A, Chu T, Mitchell JR. Surgical stress resistance induced by single amino acid deprivation requires Gcn2 in mice. Sci Transl Med. 2012 Jan 25;4(118):118ra11. doi: 10.1126/scitranslmed.3002629. PMID 22277968
- [Background] Crenshaw JT, Winslow EH. Preoperative fasting: old habits die hard. Am J Nurs. 2002 May;102(5):36-44; quiz 45. doi: 10.1097/00000446-200205000-00033. PMID 12006853
- [Background] Voute MT, Winkel TA, Poldermans D. Optimal medical management around the time of surgery. Heart. 2010 Nov;96(22):1842-8. doi: 10.1136/hrt.2008.151480. No abstract available. PMID 20965994
- [Background] Aksungar FB, Topkaya AE, Akyildiz M. Interleukin-6, C-reactive protein and biochemical parameters during prolonged intermittent fasting. Ann Nutr Metab. 2007;51(1):88-95. doi: 10.1159/000100954. Epub 2007 Mar 19. PMID 17374948
- [Background] Wycherley TP, Brinkworth GD, Noakes M, Buckley JD, Clifton PM. Effect of caloric restriction with and without exercise training on oxidative stress and endothelial function in obese subjects with type 2 diabetes. Diabetes Obes Metab. 2008 Nov;10(11):1062-73. doi: 10.1111/j.1463-1326.2008.00863.x. Epub 2008 Apr 22. PMID 18435772
- [Background] Ibrahim WH, Habib HM, Jarrar AH, Al Baz SA. Effect of Ramadan fasting on markers of oxidative stress and serum biochemical markers of cellular damage in healthy subjects. Ann Nutr Metab. 2008;53(3-4):175-81. doi: 10.1159/000172979. Epub 2008 Nov 14. PMID 19011280
- [Background] Pratley RE, Coon PJ, Rogus EM, Goldberg AP. Effects of weight loss on norepinephrine and insulin levels in obese older men. Metabolism. 1995 Apr;44(4):438-44. doi: 10.1016/0026-0495(95)90049-7. PMID 7723665
- [Background] Van Nieuwenhove Y, Dambrauskas Z, Campillo-Soto A, van Dielen F, Wiezer R, Janssen I, Kramer M, Thorell A. Preoperative very low-calorie diet and operative outcome after laparoscopic gastric bypass: a randomized multicenter study. Arch Surg. 2011 Nov;146(11):1300-5. doi: 10.1001/archsurg.2011.273. PMID 22106323
- [Background] van Ginhoven TM, de Bruin RW, Timmermans M, Mitchell JR, Hoeijmakers JH, Ijzermans JN. Pre-operative dietary restriction is feasible in live-kidney donors. Clin Transplant. 2011 May-Jun;25(3):486-94. doi: 10.1111/j.1399-0012.2010.01313.x. Epub 2010 Aug 16. PMID 20718826
- [Background] Jongbloed F, de Bruin RW, Klaassen RA, Beekhof P, van Steeg H, Dor FJ, van der Harst E, Dolle ME, IJzermans JN. Short-Term Preoperative Calorie and Protein Restriction Is Feasible in Healthy Kidney Donors and Morbidly Obese Patients Scheduled for Surgery. Nutrients. 2016 May 20;8(5):306. doi: 10.3390/nu8050306. PMID 27213441
- [Background] Grundmann F, Muller RU, Reppenhorst A, Hulswitt L, Spath MR, Kubacki T, Scherner M, Faust M, Becker I, Wahlers T, Schermer B, Benzing T, Burst V. Preoperative Short-Term Calorie Restriction for Prevention of Acute Kidney Injury After Cardiac Surgery: A Randomized, Controlled, Open-Label, Pilot Trial. J Am Heart Assoc. 2018 Mar 13;7(6):e008181. doi: 10.1161/JAHA.117.008181. PMID 29535139
- [Background] Trocha KM, Kip P, Tao M, MacArthur MR, Trevino-Villarreal JH, Longchamp A, Toussaint W, Lambrecht BN, de Vries MR, Quax PHA, Mitchell JR, Ozaki CK. Short-term preoperative protein restriction attenuates vein graft disease via induction of cystathionine gamma-lyase. Cardiovasc Res. 2020 Feb 1;116(2):416-428. doi: 10.1093/cvr/cvz086. PMID 30924866
- [Background] Robertson LT, Mitchell JR. Benefits of short-term dietary restriction in mammals. Exp Gerontol. 2013 Oct;48(10):1043-8. doi: 10.1016/j.exger.2013.01.009. Epub 2013 Feb 1. PMID 23376627
- [Background] Benotti P, Blackburn GL. Protein and caloric or macronutrient metabolic management of the critically ill patient. Crit Care Med. 1979 Dec;7(12):520-5. doi: 10.1097/00003246-197912000-00002. PMID 116801
- [Background] Verweij M, van Ginhoven TM, Mitchell JR, Sluiter W, van den Engel S, Roest HP, Torabi E, Ijzermans JN, Hoeijmakers JH, de Bruin RW. Preoperative fasting protects mice against hepatic ischemia/reperfusion injury: mechanisms and effects on liver regeneration. Liver Transpl. 2011 Jun;17(6):695-704. doi: 10.1002/lt.22243. PMID 21618690
- [Background] Yu P, Nguyen BT, Tao M, Jiang T, Ozaki CK. Diet-induced obesity drives negative mouse vein graft wall remodeling. J Vasc Surg. 2014 Jun;59(6):1670-6. doi: 10.1016/j.jvs.2013.05.033. Epub 2013 Jul 19. PMID 23876511
- [Background] Nguyen BT, Yu P, Tao M, Hao S, Jiang T, Ozaki CK. Perivascular innate immune events modulate early murine vein graft adaptations. J Vasc Surg. 2013 Feb;57(2):486-492.e2. doi: 10.1016/j.jvs.2012.07.007. Epub 2012 Nov 3. PMID 23127978
- [Background] Sharma G, Tao M, Ding K, Yu D, King W, Deyneko G, Wang X, Longchamp A, Schoen FJ, Ozaki CK, Semel ME. Perivascular adipose adiponectin correlates with symptom status of patients undergoing carotid endarterectomy. Stroke. 2015 Jun;46(6):1696-9. doi: 10.1161/STROKEAHA.114.008468. Epub 2015 May 12. PMID 25967575
- [Background] Ho KJ, Xue H, Mauro CR, Nguyen B, Yu P, Tao M, Seidman MA, Brunelli SM, Ozaki CK. Impact of uremia on human adipose tissue phenotype. J Surg Res. 2013 Jan;179(1):175-82. doi: 10.1016/j.jss.2012.08.043. Epub 2012 Sep 6. PMID 23058473
- [Background] Mauro CR, Ilonzo G, Nguyen BT, Yu P, Tao M, Gao I, Seidman MA, Nguyen LL, Ozaki CK. Attenuated adiposopathy in perivascular adipose tissue compared with subcutaneous human adipose tissue. Am J Surg. 2013 Aug;206(2):241-4. doi: 10.1016/j.amjsurg.2012.07.032. Epub 2013 Jan 23. PMID 23352378
- [Background] Mauro CR, Nguyen BT, Yu P, Tao M, Gao I, Seidman MA, Nguyen LL, Ozaki CK. Inflammatory "adiposopathy" in major amputation patients. Ann Vasc Surg. 2013 Apr;27(3):346-52. doi: 10.1016/j.avsg.2012.07.017. PMID 23498310
- [Background] Yu P, Nguyen BT, Tao M, Campagna C, Ozaki CK. Rationale and practical techniques for mouse models of early vein graft adaptations. J Vasc Surg. 2010 Aug;52(2):444-52. doi: 10.1016/j.jvs.2010.03.048. Epub 2010 Jun 22. PMID 20573477
- [Background] Yu P, Nguyen BT, Tao M, Bai Y, Ozaki CK. Mouse vein graft hemodynamic manipulations to enhance experimental utility. Am J Pathol. 2011 Jun;178(6):2910-9. doi: 10.1016/j.ajpath.2011.02.014. PMID 21641408
- [Background] Yu P, Nguyen BT, Tao M, Jiang T, Mauro CR, Wang Y, Ozaki CK. Lack of interleukin-1 signaling results in perturbed early vein graft wall adaptations. Surgery. 2013 Jan;153(1):63-9. doi: 10.1016/j.surg.2012.06.005. Epub 2012 Jul 31. PMID 22853857
- [Background] Tao M, Mauro CR, Yu P, Favreau JT, Nguyen B, Gaudette GR, Ozaki CK. A simplified murine intimal hyperplasia model founded on a focal carotid stenosis. Am J Pathol. 2013 Jan;182(1):277-87. doi: 10.1016/j.ajpath.2012.10.002. Epub 2012 Nov 15. PMID 23159527
- [Background] Tao M, Yu P, Nguyen BT, Mizrahi B, Savion N, Kolodgie FD, Virmani R, Hao S, Ozaki CK, Schneiderman J. Locally applied leptin induces regional aortic wall degeneration preceding aneurysm formation in apolipoprotein E-deficient mice. Arterioscler Thromb Vasc Biol. 2013 Feb;33(2):311-20. doi: 10.1161/ATVBAHA.112.300543. Epub 2012 Dec 6. PMID 23220275
- [Background] Chan MR, Young HN, Becker YT, Yevzlin AS. Obesity as a predictor of vascular access outcomes: analysis of the USRDS DMMS Wave II study. Semin Dial. 2008 May-Jun;21(3):274-9. doi: 10.1111/j.1525-139X.2008.00434.x. Epub 2008 Apr 6. PMID 18397205
- [Background] Wong AP, Nili N, Jackson ZS, Qiang B, Leong-Poi H, Jaffe R, Raanani E, Connelly PW, Sparkes JD, Strauss BH. Expansive remodeling in venous bypass grafts: novel implications for vein graft disease. Atherosclerosis. 2008 Feb;196(2):580-9. doi: 10.1016/j.atherosclerosis.2007.06.029. Epub 2007 Aug 10. PMID 17692852